CLINICAL TRIAL: NCT01537328
Title: Progressive Rehabilitation Following Total Knee Arthroplasty
Acronym: PROG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 10-1188; R01HD065900 (NIH)
Record Dates: First submitted 2011-08-26; First posted 2012-02-23 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Osteoarthritis
Keywords: Total knee arthroplasty; quadriceps; muscle; arthroplasty; joint diseases; musculoskeletal diseases
MeSH Terms: conditions — Osteoarthritis; Joint Diseases; Musculoskeletal Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Progressive Treatment (Experimental): Progressive intervention will involve the early initiation of intensive rehabilitation using progressive exercise and faster progression to functional strengthening exercises.
  Interventions: Other: Total knee replacement rehabilitation
- Traditional treatment (Active Comparator): Traditional intervention represents the synthesis of previously published total knee arthroplasty rehabilitation programs.
  Interventions: Other: Total knee replacement rehabilitation

INTERVENTIONS:
Other: Total knee replacement rehabilitation — After total knee arthroplasty, patients will be assigned to an outpatient rehabilitation clinic, based upon geography. Patients will be enrolled randomly into one of two rehabilitation programs (PROG or TRAD). Both rehabilitation programs will take place over 12 weeks. Both groups will receive treatment for range of motion, activities of daily living and gait training, as well as a home exercise program.

SUMMARY:
The purpose of this study is to evaluate the effectiveness of a progressive resistance rehabilitation program (PROG) after total knee arthroplasty (TKA) compared to a traditional rehabilitation program (TRAD).

The investigators hypothesized:

* PROG will result in greater improvements in functional outcome measures such as: stair climbing test (SCT), timed-up-and-go test (TUG), six minute walk test (6MW), the Knee Injury and Osteoarthritis Outcome Survey (WOMAC), and knee range of motion (ROM).
* PROG will result in greater improvements in quadriceps muscle strength gains after TKA compared to TRAD.
* PROG will result in greater improvements in muscle mass and central activation compared to TRAD.

DETAILED DESCRIPTION:
Over 500,000 total knee arthroplasties (TKAs) are performed each year in the United States to alleviate pain and disability associated with knee osteoarthritis (OA), and this number is expected to grow to 3.48 million per year by the year 2030. TKA reduces pain and improves self-reported function compared to pre-operative levels, but post-operative deficits in walking speed (20% slower) and stair climbing speed (50% slower) can persist for years. Stair climbing performance is the single largest residual deficit after TKA with seventy-five percent of TKA patients reporting difficulty negotiating stairs after surgery. Collectively, these findings suggest that current rehabilitation does not adequately target the impairments that lead to long-term deficits in functional mobility after TKA.

The aim of the proposed trial is to evaluate the effectiveness of a progressive resistance rehabilitation program (PROG) after TKA compared to a traditional rehabilitation program (TRAD). The PROG intervention will involve intensive rehabilitation using progressive resistance exercise and faster progression to functional strengthening exercises. The TRAD intervention represents the synthesis of previously published TKA rehabilitation programs. Our preliminary data suggest that the PROG intervention has low risk and results in improved functional mobility and muscle strength. The investigators will measure function and strength at six time points (pre-op; 1, 2, 3, 6, and 12 months after TKA). The investigators will also evaluate the contribution of changes in muscle mass (atrophy/hypertrophy) and central activation to changes in muscle strength following PROG and TRAD interventions.

ELIGIBILITY:
Inclusion Criteria:

* undergoing a primary, unilateral knee arthroplasty
* body mass index < 40 kg/m2

Exclusion Criteria:

* severe contralateral leg OA (< 5/10 pain with stair climbing) or other unstable orthopaedic conditions that limit function
* neurological conditions that affect muscle function
* vascular or cardiac problems that limit function
* uncontrolled diabetes
* pregnancy

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2011-07; Primary Completion 2016-05 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Stair climbing test (SCT) | pre operatively (average of two weeks before surgery), change from baseline at 1, 2, 3, 6 and 12 months
  Time to ascend and descend one flight of stairs

SECONDARY OUTCOMES:
Change from baseline in Timed-up-and-go Test (TUG) | pre operatively (average of two weeks before surgery), change from baseline at 1, 2, 3, 6 and 12 months
Change from baseline in 6-minute walk test (6MW) | pre operatively (average of two weeks before surgery), change from baseline at 1, 2, 3, 6 and 12 months
Change from baseline in muscle strength | pre operatively (average of two weeks before surgery), change from baseline at 1, 2, 3, 6 and 12 months
  Isometric quadriceps and hamstrings strength.
Change from baseline in self-reported health status | pre operatively (average of two weeks before surgery), change from baseline at 1, 2, 3, 6 and 12 months
  WOMAC and SF-12
Change from baseline in muscle activation | pre operatively (average of two weeks before surgery), change from baseline at 1, 2, 3, 6 and 12 months
  Doublet interpolation for quadriceps activation.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Stevens-Lapsley, MPT, PHD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Aurora, Colorado, United States

REFERENCES:
- [Derived] Bade M, Struessel T, Paxton R, Winters J, Baym C, Stevens-Lapsley J. Performance on a Clinical Quadriceps Activation Battery Is Related to a Laboratory Measure of Activation and Recovery After Total Knee Arthroplasty. Arch Phys Med Rehabil. 2018 Jan;99(1):99-106. doi: 10.1016/j.apmr.2017.07.013. Epub 2017 Aug 31. PMID 28864244
- [Derived] Bade MJ, Struessel T, Dayton M, Foran J, Kim RH, Miner T, Wolfe P, Kohrt WM, Dennis D, Stevens-Lapsley JE. Early High-Intensity Versus Low-Intensity Rehabilitation After Total Knee Arthroplasty: A Randomized Controlled Trial. Arthritis Care Res (Hoboken). 2017 Sep;69(9):1360-1368. doi: 10.1002/acr.23139. Epub 2017 Aug 13. PMID 27813347